CLINICAL TRIAL: NCT06569134
Title: Identification of Neuroprognostic Factors for Out-of-hospital Cardiopulmonary Arrest in the North Finistère Population: Derivation and Validation of a Predictive Score
Brief Title: Identification of Neuroprognostic Factors for Out-of-hospital Cardiopulmonary Arrest (MIRA29)
Acronym: MIRA29
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0114 - MIRA29
Record Dates: First submitted 2024-08-08; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Arrest; Neurologic Dysfunction; Cognitive Impairment
MeSH Terms: conditions — Heart Arrest; Neurologic Manifestations; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
From the informatized prehospital care registry, data will be collected anonymously for all patients' requiring cardiopulmonary resuscitation for an out-of-hospital cardiac arrest within the Norther Finistere sanitary region.

First step of the model derivation will consist in multivariate analysis to extract the most pertinent variates associated with neurological outcome (evaluated using the CPC Score); Second step will consist in the use of artificial intelligence and machine-learning to derive the most discriminant score.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest requiring cardiopulmonary resuscitation

Exclusion Criteria:

* Death before cardiopulmonary resuscitation
* Pediatric Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting a cardiac arrest requiring cardiopulmonary resuscitation, taken in charge by the Northern Finistere Prehospital Care System, will be included Datafiles will be individually revised
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-07-24 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2025-01-24 (Estimated)

PRIMARY OUTCOMES:
Cognitive Outcome | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  It will be evaluated at the end of the ICU stay using the CPC score; a CPC score equal or below 2 will be considered as a good outcome, while a CPC > 2 will be considered as a bad outcome

SECONDARY OUTCOMES:
Death OoH | Before hospital arrival
  Death after resuscitation during the prehospital care phase
Death ICU | During ICU stay
  Death within the ICU care
Death at Day 28 | 28 days after cardiac arrest
  Death at Day 28, before or after hospital discharge

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Brest, Brest
  - CH des pays de Morlaix, Morlaix